CLINICAL TRIAL: NCT01675934
Title: Right-sided Retroflexion With Standard Adult Versus Pediatric Colonoscopes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has left institution
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO00017208
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Colonic Neoplasms
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adult colonoscope (Active Comparator): Use of the adult colonoscope.
  Interventions: Procedure: Retroflexion with the adult colonoscope.
- Pediatric colonoscope (Active Comparator): Use of the pediatric colonoscope.
  Interventions: Procedure: Retroflexion with the pediatric colonoscope.

INTERVENTIONS:
Procedure: Retroflexion with the adult colonoscope.
  Arms: Adult colonoscope
Procedure: Retroflexion with the pediatric colonoscope.
  Arms: Pediatric colonoscope

SUMMARY:
Screening colonoscopy has been shown to be less effective in preventing colorectal cancer in the proximal colon compared to the distal colon. Possible reasons for this include bowel preparation often being worse in the proximal colon as well as flat depressed lesions being more common in the proximal colon.

Retroflexion is commonly regarded as standard practice in the rectum, but retroflexion in the proximal colon is not currently routinely performed due to concerns of perforation and possibly because of the increased time required.

Proximal colon retroflexion has been shown to be safe and effective without any complications, but data regarding ability to retroflex with certain types of colonoscopes is limited. Endoscopists interchangeably use standard adult colonoscopes or pediatric colonoscopes. Studies have not been performed to comparatively evaluate the success rates of standard adult and pediatric colonoscopes and whether either type of instrument confers a greater polyp detection rate.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over the age 18 undergoing screening or surveillance colonoscopy

Exclusion Criteria:

* Age less than 18
* Pregnant
* History of ulcerative colitis or Crohn's disease
* History of polyposis syndromes
* History of colon resection
* Colonoscopy being performed for diagnostic purposes (ie. bleeding, abdominal pain, alternating bowel habits)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Percentage of cases in which right-sided retroflexion is successful with the adult and pediatric colonoscopes. | After 50% and 100% of patient enrollment is complete.

SECONDARY OUTCOMES:
Adenoma detection rate in forward and retroflexed views. | After 50% and 100% of patient enrollment is complete.
Reasons for failure of retroflexion. | After 50% and 100% of patient enrollment is complete.
  This will be assessed as a yes/no variable. In addition, the specific reasons that the endoscopist could not retroflex the colonoscope in the right colon will assessed, such as the colonoscope not being able to be advanced to the cecum, small diameter of the right colon, too much resistance encountered when attempting retroflexion that the endoscopist does not feel comfortable with, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Young Oh, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Surgery Center, Milwaukee, Wisconsin, United States